CLINICAL TRIAL: NCT01563653
Title: Development and Evaluation of a New Diagnostic Test in Female Urinary Stress Incontinence
Acronym: IEUF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough inclusions.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2011/RdeT-01; 2011-A01225-36 (Other: RCB number)
Record Dates: First submitted 2012-03-16; First posted 2012-03-27 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Urinary Incontinence, Stress
Keywords: predicting surgical success; simple diagnostic test device
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Women with stress urinary incontinence schelduled for TVT or TOT procedures. See inclusion/exclusion criteria.
  Interventions: Procedure: 4 diagnostic tests for surgical success

INTERVENTIONS:
Procedure: 4 diagnostic tests for surgical success — Q-tip test, Bonney maneuver, TVT maneuver, clip strip test

SUMMARY:
The investigators hypothesize that an innovative test device simulating transvaginal tape support will increase the performance and reproducibility of the diagnosis of urethral hypermobility before surgery for urinary incontinence.

The main objective of this study is to compare two prognostic tests in their ability to predict the success (or failure) of the implementation of a suburethral TVT (tension-free vaginal tape) or TOT (trans-obturator tape) treatment for stress urinary incontinence in women. The Q-tip test (test mentioned in the French and international recommendations) is compared to test a new test (clip strip).

DETAILED DESCRIPTION:
Secondary objectives include:

* Compare the prognostic ability of the clip strip test with the Bonney maneuver
* Compare the prognostic ability of the clip strip test with the TVT maneuver
* Compare the maximum intraurethral pressure during various tests
* Compare the quality of life before / after surgery
* Estimate patient satisfaction one year after surgery
* Describe the intra and inter-operator reproducibility of various prognostic tests.
* Estimate the optimal threshold of the Q-tip angle based on surgical results and compare with the reference threshold of 30 ° found in the literature.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 60 weeks of follow-up
* Candidate for stress urinary incontinence surgery by TVT or TOT procedures
* Positive cough or valsalve maneuver test

Exclusion Criteria:

* The patient is participating in another study (except the PISQ-R study)
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contra-indication for stress urinary incontinence surgery via TVT or TOT procedures.
* The patient has an untreated vaginal or urniary infection
* The patient has a history of allergy to polyurethane and / or Watershed XCX11122

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
McNemar Score: Comparison of Q-tip test and clip strip test results with surgical results | 58-60 weeks
  McNemar test for comparing sensitivity and specificity between two factors

SECONDARY OUTCOMES:
McNemar Score: Comparison of Q-tip test and clip strip test results with surgical results | 2-4 weeks
  McNemar test for comparing sensitivity and specificity between two factors
McNemar Score: Comparison of Q-tip test and clip strip test results with surgical results | 6-8 weeks
  McNemar test for comparing sensitivity and specificity between two factors
Positive Bonney maneuver | 2-4 weeks
  yes/no
Positive Bonney maneuver | 6-8 weeks
  yes/no
Positive TVT maneuver | 2-4 weeks
  yes/no
Positive TVT maneuver | 6-8 weeks
  yes/no
McNemar Score: Clip strip test versus Bonney maneuvre | 58-60 weeks
  Comparison of the prognostic capacities of the clip strip and Bonney maneuver tests. McNemar test for comparing sensitivity and specificity between two factors
McNemar Score: Clip strip test TVT Bonney maneuvre | 58-60 weeks
  Comparison of the prognostic capacities of the clip strip and TVT maneuver tests. McNemar test for comparing sensitivity and specificity between two factors
Intra-urethral pressure during the Bonney maneuver | 2-4 weeks
  mm Hg
Intra-urethral pressure during the Bonney maneuver | 6-8 weeks
  mm Hg
Intra-urethral pressure during the TVT maneuver | 6-8 weeks
  mm Hg
Intra-urethral pressure during the TVT maneuver | 2-4 weeks
  mm Hg
Intra-urethral pressure during the clip strip test | 2-4 weeks
  mm Hg
Intra-urethral pressure during the clip strip test | 6-8 weeks
  mm Hg
UDI-6 questionnaire | 2-4 weeks
UDI-6 questionnaire | 12-14 weeks
UDI-6 questionnaire | 58-60 weeks
IIQ7 questionnaire | 2-4 weeks
IIQ7 questionnaire | 12-14 weeks
IIQ7 questionnaire | 58-60 weeks
PGI-I Questionnaire | 58-60 weeks
Intra- and inter operator reproducability for 4 diagnostic tests | 2-4 weeks
  Bonney maneuver, q-tip test, tvt maneuver and clip strip test
Intra- and inter operator reproducability for 4 diagnostic tests | 6-8 weeks
  Bonney maneuver, q-tip test, tvt maneuver and clip strip test
Angle associated with Q-tip test | 2-4 weeks
Angle associated with Q-tip test | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Renaud de Tayrac, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - CH de Dignes les Bains, Digne-les-Bains